CLINICAL TRIAL: NCT00368498
Title: A Randomized Single Blind Parallel Control Trial to Evaluate the Loading Dose Required to Achieve Therapeutic Serum Teicoplanin Concentration Timely
Brief Title: A Trial to Evaluate the Loading Dose Required to Achieve Therapeutic Serum Teicoplanin Concentration Timely
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 950115
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2006-08-24 (Estimated); Status verified 2006-08

CONDITIONS: Staphylococcal Infections
Keywords: teicoplanin
MeSH Terms: conditions — Staphylococcal Infections | interventions — Teicoplanin

INTERVENTIONS:
Drug: teicoplanin

SUMMARY:
The purpose of this study is to determine whether the standard dosage of teicoplanin is adequate to produce timely the trough level > 10 mg/L, which is considered to be effective in the treatment of methicillin-resistant Staphyllococcus aureus (MRSA) bacteremia.

DETAILED DESCRIPTION:
In our hospital, the minimum inhibitory concentration of 100 MRSA isolates in 2003 for teicoplanin is 2 mg/L. Due to its time-dependant bacteriocidal effect, the trough level should exceed 10 mg/L, particularly in the elderly, for MRSA bacteremia. However, it is known that standard dosage of teicoplanin often produces inadequate serum trough levels, and MRSA infections may recurred. Therefore, to evaluate the loading dose required to achieve therapeutic concentration timely, we compare the trough levels between those given standard dose (6 mg/Kg) and those given increasing loading dose (12 mg/Kg). We also monitor the occurrence of adverse drug effects and clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 16 years of age who have blood culture-proven MRSA bacteremia and did not receive teicoplanin or vancomycin in the previous one month are enrolled.

Exclusion Criteria:

* Those who are allergic to teicoplanin or who have the need to use higher doses, 12 mg/kg/dose, such as endocarditis, osteomyelitis, septic arthritis and burn patients, are excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2006-06; Study Completion 2007-12

PRIMARY OUTCOMES:
the proportion of the trough level attaining 10 mg/L at different timing

SECONDARY OUTCOMES:
the occurrence of adverse drug effects
the correlation between the trough level and the patients' characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Shan-Chwen Chang, Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan